CLINICAL TRIAL: NCT07139821
Title: Dietary Iron Requirements in US Adults
Brief Title: Dietary Iron Requirements
Status: Not yet recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-036-PBRC
Record Dates: First submitted 2025-08-07; First posted 2025-08-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Iron Absorption
Keywords: Iron absorption; Iron losses; Iron requirements; Iron deficiency; Iron deficiency anemia; Iron isotopes
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- US adult males and premenopausal females: A representative sample of adult males and premenopausal females living in the US

SUMMARY:
Dietary Reference Intakes (DRIs) for iron are based on a relatively small number of studies in European populations. This research study will determine iron needs in a representative sample of adults living in the US using the iron isotope dilution technique. Following administration and equilibration of a stable iron isotope, participants will be followed for a 12 week study period. Blood will be collected every 4 weeks and the isotopic composition will be determined. Results will help update dietary iron guidelines making sure they better match the specific needs of the US population.

ELIGIBILITY:
Inclusion Criteria:

* Males and premenopausal females age 18-50 y
* Previously participated in an iron stable isotope study or willing to consume an oral stable iron isotope and undergo a one-year equilibration period
* Willing to refrain from iron-containing supplements for the duration of the study
* Willing to refrain from tobacco smoking for the duration of the study
* Have not donated blood 3 months prior to the start of the study and willing to refrain from donating blood for the duration of the study
* Willing to have blood stored for future use
* Able and willing to comply with study requirements and consent to participate

Exclusion Criteria:

* Females: pregnant or lactating or plans to become pregnant during the study period
* Inability to provide informed consent and engage in informed consent procedures
* Plans to relocate outside the study area

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be enrolled at LSU Pennington Biomedical Research Center in Baton Rouge, Louisiana and Cornell University in Ithaca, New York.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Iron isotope composition in blood | 12 weeks
  Tracer-to-tracee rate in venous blood samples collected at multiple time points

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - LSU Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Cornell University, Ithaca, New York

IPD SHARING:
Plan to Share IPD: No